CLINICAL TRIAL: NCT02373215
Title: A Phase 1, Open-Label, Non-Randomized, Parallel-Group Study to Characterize and Compare the Pharmacokinetics, Safety, and Tolerability of Escalating Oral Doses of Nalbuphine Hydrochloride Extended Release Tablets in End-Stage Renal Disease Patients on Hemodialysis and Matched Healthy Control Subjects
Brief Title: Phase 1 Study of Nalbuphine HCl ER Tablets in Hemodialysis Patients With Uremic Pruritus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR01
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Uremic Pruritus
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 - Groups 1-3 (Experimental): HD patients dosing up to 180mg BID
  Interventions: Drug: Nalbuphine HCL ER
- Cohort 1 - Group 4 (Experimental): HD patients dosing up to 240mg BID
  Interventions: Drug: Nalbuphine HCL ER
- Cohort 2 (Experimental): Healthy patients dosing up to 180mg BID
  Interventions: Drug: Nalbuphine HCL ER

INTERVENTIONS:
Drug: Nalbuphine HCL ER — Nalbuphine HCL extended release tablet
  Other Names: Nalbuphine

SUMMARY:
This is a single-center clinical research study with the purpose to evaluate the safety, tolerability, and pharmacokinetics (PK) of nalbuphine HCl ER (extended release) tablets in end-stage renal disease (ESRD) patients receiving hemodialysis (HD) therapy and reporting pruritus.

DETAILED DESCRIPTION:
The PK of nalbuphine hemodialysis (HD) patients is unknown and will be investigated under controlled dialysis conditions in the proposed clinical PK study.

Nalbuphine is a small molecular weight, water-soluble molecule with low protein binding (approximately 50%) and a large volume of distribution. In addition, its disposition is perfusion-rate limited. In the end-stage renal disease (ESRD) patients on HD, nalbuphine plasma clearance may be impacted, although it is predominantly hepatically cleared in the feces.

A dose-escalation design was selected to mimic nalbuphine use in uremic pruritus (UP) patients in subsequent clinical efficacy studies whereby patients will start at a low dose to minimize the AEs such as nausea and vomiting and allow the patients to develop some tolerance to these particular AEs.

ELIGIBILITY:
Inclusion Criteria:

For Hemodialysis Patients Only

1. Patients with chronic renal failure who have been receiving chronic in-center HD on an average of 3 times a week for at least 3 months (with Kt/V > 1.1).
2. Subjects who experience at least mild intermittent pruritus.
3. Non-reactive serology for hepatitis B, hepatitis C, and human immunodeficiency virus (HIV) antibody screens.
4. Adequate venous access.
5. Hemoglobin concentration at Screening > 9 g/dL.

For Healthy Subjects Only

1. Subjects are demographically comparable to the ESRD subjects.

   1. Gender matched 100%
   2. Age ± 10 years
   3. Body mass index (BMI) ± 15%
2. Clinical chemistry within normal range.

For Hemodialysis Patients and Healthy Subjects

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female between the ages of 18 and 70 years, inclusive.

Exclusion Criteria:

For Hemodialysis Patients Only

1. Patients who had a significant alteration in dialysis regimen within 2 weeks of the Screening Visit.
2. An alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) concentration > 2x the upper limit of the normal range (ULN) at Screening.
3. A serum total bilirubin > 1.8x ULN.
4. Patients who require peritoneal dialysis.
5. Patients who received daily or when necessary (PRN) barbiturates, amphetamines, or opiates within 7 days prior to Check-in.

For Healthy Subjects Only

1. Any clinically significant abnormality identified on the physical, ECG, vital sign measurements, or clinical laboratory examinations at Screening or Day -1.

For Hemodialysis Patients and Healthy Subjects

1. Subjects with a positive drug screen at Screening and Day -1 without a prescription.
2. Known hypersensitivity or allergy to nalbuphine or vehicle components.
3. Known drug allergy to opioids.
4. History of drug dependency, opioid abuse, or emotional instability deemed clinically significant per investigator review.
5. Women with a positive pregnancy test
6. Lactating females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Steady state PK of nalbuphine HCl ER tablets as a function of dose | Day -1 to 14 Cohort 1 Groups 1-3 and Cohort 2; Day -1 to 17 Cohort 1 Group 4
  Steady state PK of nalbuphine HCl ER tablets following escalating repeated oral doses in ESRD patients receiving HD therapy relative to healthy subjects
Extent of extraction of nalbuphine by measuring nalbuphine in plasma and dialysate during dialysis | Day -1 to 14 Cohort 1 Groups 1-3; Day -1 to 17 Cohort 1 Group 4
  Extraction by dialysis was assessed by measuring nalbuphine concentrations in plasma during dialysis obtained from arterial (pre-dialyzer) and venous access ports (post-dialyzer) and by measuring the amount removed in the dialysate during dialysis in the dialysate as a function of dose.

SECONDARY OUTCOMES:
VAS measurement of anti-pruritic effects | Day -1 to 19-21 Cohort 1 Groups 1-3; Day -1 to 22-24 Cohort 1 Group 4
  Visual Analogue Scale (VAS) itch measurement of anti-pruritic effects of nalbuphine HCl ER tablets in HD subjects with pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics

REFERENCES:
- [Derived] Eudy-Byrne R, Riggs M, Hawi A, Sciascia T, Rohatagi S. A population pharmacokinetic-pharmacodynamic model evaluating efficacy of nalbuphine extended-release in patients with prurigo nodularis. Br J Clin Pharmacol. 2023 Jul;89(7):2088-2101. doi: 10.1111/bcp.15663. Epub 2023 Feb 9. PMID 36680419